CLINICAL TRIAL: NCT05898945
Title: Primary Repair of Obstetric Anal Sphincter Injuries (OASIS): a Survey of Emergency Surgeons' Experience
Brief Title: Primary Repair of Obstetric Anal Sphincter Injuries (OASIS) by Surgeons (PROS Study)
Acronym: PROS
Status: Completed | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 326703
Record Dates: First submitted 2023-03-15; First posted 2023-06-12 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-06

CONDITIONS: Obstetric Anal Sphincter Injury
Keywords: primary repair; management; emergency surgeons; incontinence; outcomes; survey; coloproctologists

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Third- or fourth-degree perineal tears, collectively known as Obstetric Anal Sphincter Injuries or OASIS, may occur following a vaginal birth. OASIS may have catastrophic consequences, including anal incontinence. Satisfactory primary repair of OASIS is prudent in reducing the risk of maternal morbidity. Although Obstetricians are typically involved in the acute repair of OASIS, General Surgeons may be called to assist in cases of severe anatomical disruption.

The investigators have constructed a survey to explore the experience and current practice of Emergency Surgeons in relation to the repair of OASIS. The investigators will gather information including their level of exposure, understanding of current guidelines and confidence in performing these repairs. This will help the investigators identify if further training is required and will enable them to put forward recommendations for future practice. The findings will be presented at conferences and meetings and published in journals.

DETAILED DESCRIPTION:
To date, there is little consensus on who should perform the primary repair of obstetric anal sphincter injuries (OASIS), with the Royal College of Obstetricians and Gynaecologists (RCOG) stating that the repair should be undertaken by a trained practitioner and that 'involvement of a colorectal surgeon will be dependent on local protocols, expertise and availability'.

In cases of severe anatomical disruption, the on-call general surgeon may be summoned upon to assist with the repair. They may not be a colorectal surgeon, and if they are, they may not specialise in pelvic floor surgery. A previous survey of practice amongst UK obstetricians and coloproctologists identified a wide variation in experience, methods of repair, follow up and recommendations for future delivery.

The aim of this study is to explore emergency surgeons' knowledge in relation to the acute repair of OASIS and to compare this with current recommendations and best practice guidance. This, in turn, will help identify if further training is required.

Satisfactory repair of acute OASIS is necessary for the following reasons:

* It may reduce the risk of anal incontinence, a stigmatising condition which may have substantial impact on an individual's quality of life and day-to-day living.
* By reducing the incidence of OASIS-related anal incontinence, the financial burden associated with the management of this condition as well as the risk of litigation will also be reduced

ELIGIBILITY:
Inclusion Criteria:

* Registrar or above
* Cover an Emergency on-call rota for General Surgery
* Working in Great Britain and Ireland

Exclusion Criteria:

* • Senior House Officers or Foundation Doctors

  * Doctors who do not cover an emergency rota
  * Doctors working abroad

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency general surgeons (registrar or consultant level) are eligible to participate. This includes registrar trainees (StR), staff grades, associate specialists, speciality doctors and consultants who are on the speciality register. They will need to be participating in an emergency on-call rota and working in Great Britain and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Use of Knowledge | study to be completed over a 12 month period
  Ascertainment of the knowledge of trainee, SAS and consultant (varying in age, sub-speciality and region) knowledge and skills in primary OASI repairs, in guideline and policy-related documents and adherence to management recommendations, using a questionnaire
Training and confidence | study to be completed over a 12 month period
  Effect of the number of OASI repairs performed throughout the career of trainees, SAS and consultants (varying in age, sub-speciality and region) and training received, on confidence in performing OASI repairs, using a questionnaire

SECONDARY OUTCOMES:
Knowledge-related attitudes | study to be completed over a 12 month period
  Accurate mapping of the pathway of patient follow-up processes following OASI repairs, using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- London North West University Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurol-Urganci I, Cromwell DA, Edozien LC, Mahmood TA, Adams EJ, Richmond DH, Templeton A, van der Meulen JH. Third- and fourth-degree perineal tears among primiparous women in England between 2000 and 2012: time trends and risk factors. BJOG. 2013 Nov;120(12):1516-25. doi: 10.1111/1471-0528.12363. Epub 2013 Jul 3. PMID 23834484
- [Background] Bols EM, Hendriks EJ, Berghmans BC, Baeten CG, Nijhuis JG, de Bie RA. A systematic review of etiological factors for postpartum fecal incontinence. Acta Obstet Gynecol Scand. 2010 Mar;89(3):302-14. doi: 10.3109/00016340903576004. PMID 20199348
- [Background] Snooks SJ, Setchell M, Swash M, Henry MM. Injury to innervation of pelvic floor sphincter musculature in childbirth. Lancet. 1984 Sep 8;2(8402):546-50. doi: 10.1016/s0140-6736(84)90766-9. PMID 6147604
- [Background] Sioutis D, Thakar R, Sultan AH. Overdiagnosis and rising rate of obstetric anal sphincter injuries (OASIS): time for reappraisal. Ultrasound Obstet Gynecol. 2017 Nov;50(5):642-647. doi: 10.1002/uog.17306. PMID 27643513
- [Background] Andrews V, Sultan AH, Thakar R, Jones PW. Occult anal sphincter injuries--myth or reality? BJOG. 2006 Feb;113(2):195-200. doi: 10.1111/j.1471-0528.2006.00799.x. PMID 16411998
- [Background] Abramov Y, Feiner B, Rosen T, Bardichev M, Gutterman E, Lissak A, Auslander R. Primary repair of advanced obstetric anal sphincter tears: should it be performed by the overlapping sphincteroplasty technique? Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1071-4. doi: 10.1007/s00192-008-0592-0. Epub 2008 Apr 3. PMID 18385917
- [Background] Fernando R, Sultan AH, Kettle C, Thakar R, Radley S. Methods of repair for obstetric anal sphincter injury. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD002866. doi: 10.1002/14651858.CD002866.pub2. PMID 16855993
- [Background] Fernando RJ, Sultan AH, Radley S, Jones PW, Johanson RB. Management of obstetric anal sphincter injury: a systematic review & national practice survey. BMC Health Serv Res. 2002 May 13;2(1):9. doi: 10.1186/1472-6963-2-9. PMID 12006105
- [Background] Sultan AH, Kamm MA, Hudson CN, Bartram CI. Third degree obstetric anal sphincter tears: risk factors and outcome of primary repair. BMJ. 1994 Apr 2;308(6933):887-91. doi: 10.1136/bmj.308.6933.887. PMID 8173367
- [Background] Norderval S, Markskog A, Rossaak K, Vonen B. Correlation between anal sphincter defects and anal incontinence following obstetric sphincter tears: assessment using scoring systems for sonographic classification of defects. Ultrasound Obstet Gynecol. 2008 Jan;31(1):78-84. doi: 10.1002/uog.5155. PMID 18059077